CLINICAL TRIAL: NCT03910452
Title: Haploidentical Transplant for Patients With Chronic Granulomatous Disease (CGD) Using Alemtuzumab, Busulfan and TBI With Post-Transplant Cyclophosphamide
Brief Title: Haploidentical Transplant for People With Chronic Granulomatous Disease (CGD) Using Alemtuzumab, Busulfan and TBI With Post-Transplant Cyclophosphamide
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190080; 19-I-0080
Record Dates: First submitted 2019-04-09; First posted 2019-04-10 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09-11

CONDITIONS: Chronic Granulomatous Disease
Keywords: Haplo-identical; Allogeneic Stem Cell Transplant; Peripheral Blood Stem Cell Transplant; Graft Versus Host Disease; Non-Myeloablative Conditioning Regimen
MeSH Terms: conditions — Granulomatous Disease, Chronic; Graft vs Host Disease | interventions — Busulfan; Alemtuzumab; Cyclophosphamide; Sirolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): This is a single arm open-label pilot study.
  Interventions: Drug: Busulfan; Drug: Alemtuzumab; Drug: Cyclophosphamide; Drug: Sirolimus; Radiation: Total Body Irradiation; Biological: Allogeneic peripheral blood stem cell

INTERVENTIONS:
Drug: Busulfan — 3 days of IV Busulfan. An alkylating chemotherapeutic agent determined to have broad myelosuppressive effects. On this study is being used as part of conditioning regimen for myelosuppressive properties as per package insert and standard of care.
Drug: Alemtuzumab — 5 days of IV Alemtuzumab. A humanized monoclonal antibody directed against CD52 (which is abundantly expressed on all human lymphocytes), and causes T cell activation in vitro as well as complement-mediated lysis and antibody-dependent cellular toxicity. For this study, being used as part of the conditioning regimen per package insert and standard of practice.
Drug: Cyclophosphamide — 2 days of IV Cyclophosphamide. This is an antineoplastic, and for this study is bine used for its immunosuppressive mechanism of action per package insert and standard of care
Drug: Sirolimus — Post Peripheral blood stem cell infusion. It is used for its immunosuppressive mechanism of action.
Radiation: Total Body Irradiation — 2 fractionated doses on -2 day. It is used for its immunosuppressive mechanism of action. It is SOP for conditioning for transplant.
Biological: Allogeneic peripheral blood stem cell — IV infused donor peripheral blood stem cell. Stem cells are cells that give rise to the blood cells - red blood cells that carry oxygen, white blood cells that help the body to fight infections, and platelets that help make the blood clot. Collected and infused per the standard of operating procedures established by the Department of Transfusion Medicine.

SUMMARY:
Background:

CGD causes infections and inflammation. The only cure currently is a bone marrow transplant. Most often a perfectly matched bone marrow donor is used. Researchers want to see if they can lower the risks of using a mismatched donor.

Objectives:

To see if it is safe to use a related bone marrow donor who is only a partial match to a person with CGD. To see how well drugs given to a person before and after transplant help the body accept the transplant.

Eligibility:

People ages 4-65 with CGD for whom stem cell transplant may be a cure and who do not have a perfectly matched donor, related or unrelated.

Design:

Participants will be screened with:

Medical history

Physical exam

Blood tests

Participants will be admitted to the hospital about 2 weeks before the transplant. They will have blood, urine, breathing, and heart tests. They may have CT and/or MRI scans. They will have a needle inserted into their hipbone to remove marrow. They will have dental, neurologic, and psychologic tests. They will have a central catheter placed: A line will be placed into a vein in their upper chest. They will get drugs, chemotherapy, and radiation to prepare for the transplant.

Participants will receive the donated cells through their catheter. The cells will be from one of their relatives.

Participants will stay in the hospital about 6 weeks after the transplant.

After they leave the hospital, participants will have to stay in the area with visits about 2 times a week for approximately 100 days post transplant. Then visits will be every 3 to 6 months for 2 years. Then visits will be once a year.

DETAILED DESCRIPTION:
Allogeneic transplant using human leukocyte antigen (HLA) matched donors, both related and unrelated, has proven curative for patients with various immunodeficiencies, including those with ongoing infections. However, donor availability remains a limiting factor in the application of this treatment modality. For this protocol, a haploidentical donor is a related donor with more than 1 HLA antigen mismatch. The use of haploidentical related donors has in the past been fraught with a greater rate of complications related to both higher rates of graft versus host disease (GvHD) and delayed immunorecovery. Newer transplant regimens appear to have diminished these risks and improved outcomes. We propose using a reduced intensity novel conditioning regimen using alemtuzumab, targeted busulfan, and low dose total body irradiation (see schema below) followed by post-transplant cyclophosphamide for patients with chronic granulomatous disease (CGD) who do not have an HLA matched donor but whose circumstances necessitate the use of a potentially curative, albeit high-risk treatment modality. However, patients with CGD have high rates of Crohn s Disease-like inflammatory bowel disease, predominantly colitis, where uncontrolled severe IBD may increase risk of GvHD. For this reason, the first 10 patients enrolled will exclude those deemed to have intestinal inflammation in the severe category.

As part of the study design, the protocol will enroll patients sequentially.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Must have sufficient complications from underlying disease to warrant undergoing transplantation. (History of one or more life threatening infections and/or an ongoing infection not responsive to current medical therapy and/or ongoing inflammation along with an oxidase level within quartile 1 or 2.
* Patients will be reviewed at a multidisciplinary meeting for assessment of the risk/benefit ratio of transplant for the patient to determine suitability for this high risk treatment. This multidisciplinary meeting is a combined NCI/NIAID bimonthly meeting comprised of investigators from multiple branches of the NC and NIAID to review patients with immunodeficiencies being considered for various transplant protocols.
* Patients who are deemed to have colitis in the severe category (severe colitis) as defined below in the Subject Exclusion Criteria, who are at high risk for GvHD, will be included in enrollment to the protocol after 10 patients have completed the protocol regimen successfully. Patients among the first 10 may have colitis that is not deemed in the severe category. The success of the regimen will be determined as engraftment with a maximum GvHD of grade 2 (See the exclusion criteria for patients with severe colitis).
* Patients who are 4 65 years of age.
* HLA mismatched related (more than 1 mismatch) donor graft available.
* Ability to comprehend and willingness to sign the informed consent or have a parent/guardian consent if the donor is a minor; assent being obtained from minors as appropriate.
* Must be HIV negative.
* Must be able to stay within one hour s travel of the NIH for the first 3 months after transplantation and have a family member or other designated companion to stay with during the post-transplant period.
* Must provide a durable power of attorney for health care decisions to an appropriate adult relative or guardian in accordance with NIH Form-200 NIH Durable Power of Attorney for Health Care Decision Making."
* Where appropriate, subjects must agree to use contraception for 3 months post-transplant.

NOTE: Alemtuzumab (IV formulation) is no longer distributed commercially. In order to receive product, the physician must contact the program for the patient. If the subject is not willing to consent to submit their info (address, date of birth and gender) to the program such that we can obtain the drug, then we cannot proceed with conditioning therefore no transplant will occur on this protocol.

Participation of Women:

Contraception: The effects of the combination of conditioning medications (alemtuzumab, busulfan, cyclophosphamide and mycophenolate mofetil) and total body irradiation on the developing human fetus are unknown. For this reason, men and women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for at least one year post transplant. Females of childbearing-age must have a negative pregnancy test result prior to receiving any chemotherapy or conditioning agents. During the course of the study, if a woman becomes pregnant or suspects she is pregnant, she should inform the study staff and her primary care physician immediately.

Participation of Children:

Children greater than or equal to 4 years of age may participate in this study.

EXCLUSION CRITERIA:

* The subject cannot have a 9/10 or 10/10 HLA matched related or unrelated donor.
* Eastern Cooperative Oncology Group (ECOG) or equivalent performance status greater than or equal to 3
* Patients with inflammatory bowel disease deemed in the severe category (severe colitis), because they are at higher risk for GvHD, will be excluded from the protocol until there are 10 patients without severe colitis that have successfully completed a regimen, as determined by engraftment and acute GvHD of a maximum of grade 2. Severity of colitis will be determined in consultation with a gastroenterologist specialist. However, severe colitis will be evaluated within 4 months of transplant and defined as any of the following (where this screening may be performed on a natural history or screening protocol):

  * The consultant gastroenterologist clinically determines that the patient has severe colitis.
  * Patient adult CDAI score is in the 350-450 range and Pediatric CDAI score is greater than 30 within the month before initiation of conditioning Crohn s Disease Activity Index (CDAI) for transplant.
  * The patient has been requiring 1 mg/kg/day or more of prednisone or equivalent steroid for control of colitis within 1 month of the CDAI scoring used to determine eligibility.
  * The patient requires continuing treatment with a biologic that consists of anti-TNF alpha (e.g. infliximab, Humira, certolizumab and others of this family), anti-interleukin 12 (e.g. Ustekinumab) or anti-integrin (e.g. Vedolizumab) for control of colitis within 2 months of the CDAI scoring used to determine eligibility.
  * If the patient had a colonoscopy within 6 months of transplant which revealed findings of a simplified endoscopic score of Crohn s Disease (SES-CD) greater than 15.
* Left ventricular ejection fraction < 40%.
* Transaminases > 5x upper limit of normal.
* Psychiatric disorder or mental deficiency severe enough as to make compliance with the HSCT treatment unlikely, and/or making regulatorily and legally effective informed consent impossible. This will include adult patients that are unable to consent.
* Major anticipated illness or organ failure incompatible with survival from AlloPBSC transplant.
* Pregnant or lactating.
* HIV positive.
* Participants older than 65 are excluded. It is known from standard transplantation that these participants have a higher risk of morbidity and mortality related to transplantation. Given the investigational nature of this protocol, the risk benefit ratio is not warranted to include these participants at this time.
* Participants who are not willing to submit their information as part of the alemtuzumab (Campath ) Distribution Program application or participants whom the Distribution Program committee has determined are not qualified to receive alemtuzumab.
* Any condition or circumstance, which the Principal Investigator (PI) feels, would create difficulty in maintaining compliance with the requirements of this protocol.
* Any active infectious disease, whether CGD-related or not, that is deemed to be incompatible with successful tolerance to the rigors of transplantation.
* C-reactive protein of greater than 100 Units within 6 weeks of anticipated transplant.
* Any history of seizures, controlled or otherwise, if unrelated to an infectious cause.
* Any history of any neurologic disorders or family history of such, unrelated to infection.
* Brain CT or MRI findings suggestive of neurologic disorders other than infection.

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2034-06-15 (Estimated); Study Completion 2034-06-15 (Estimated)

PRIMARY OUTCOMES:
Engraftment - Chimerism | Day 30, 100, 6mo, 12 mo
  Myeloid chimerism >50% without incurring grade 3 steroid refractory or any grade 4 acute graft versus host disease or severe extensive chronic graft versus host disease post transplant.

SECONDARY OUTCOMES:
Viral immune titrels | 6 mo, 1 year, 2 year, and 3 years post transplant.
  Viral Immune Reconstitution using viral reactivation as a marker.
Overall Survival/Event-Free survival | continuous observation/Day +14, 30, 60, 100, 6 mo, 12 mo, 18 mo, 2,3,4,5 years
  3) Assessment of rates of Overall Survival and Event Free Survival (event being late graft loss or recurrence of CGD phenotype).
DHR as a marker of normal neutrophil function | Day 30, 100, 6 month and 1 year
  1) Myeloid immune reconstitution levels with DHR as a marker of normal neutrophil function by 1-year post transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Kang, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marsh RA, Kim MO, Liu C, Bellman D, Hart L, Grimley M, Kumar A, Jodele S, Myers KC, Chandra S, Leemhuis T, Mehta PA, Bleesing JJ, Davies SM, Jordan MB, Filipovich AH. An intermediate alemtuzumab schedule reduces the incidence of mixed chimerism following reduced-intensity conditioning hematopoietic cell transplantation for hemophagocytic lymphohistiocytosis. Biol Blood Marrow Transplant. 2013 Nov;19(11):1625-31. doi: 10.1016/j.bbmt.2013.09.001. Epub 2013 Sep 10. PMID 24035782
- [Background] Munchel A, Kesserwan C, Symons HJ, Luznik L, Kasamon YL, Jones RJ, Fuchs EJ. Nonmyeloablative, HLA-haploidentical bone marrow transplantation with high dose, post-transplantation cyclophosphamide. Pediatr Rep. 2011 Jun 22;3 Suppl 2(Suppl 2):e15. doi: 10.4081/pr.2011.s2.e15. PMID 22053277
- [Background] Parta M, Kelly C, Kwatemaa N, Theobald N, Hilligoss D, Qin J, Kuhns DB, Zerbe C, Holland SM, Malech H, Kang EM. Allogeneic Reduced-Intensity Hematopoietic Stem Cell Transplantation for Chronic Granulomatous Disease: a Single-Center Prospective Trial. J Clin Immunol. 2017 Aug;37(6):548-558. doi: 10.1007/s10875-017-0422-6. Epub 2017 Jul 28. PMID 28752258
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-I-0080.html